CLINICAL TRIAL: NCT01899625
Title: Using Motivational Interviewing to Improve Weight Loss Outcomes With Young Adults
Brief Title: Motivational Interviewing for Weight Loss With Young Adults
Acronym: LiveWellRVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM14613; R03DK095959 (NIH)
Record Dates: First submitted 2013-07-06; First posted 2013-07-15 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
Keywords: Obesity; weight loss; young adults
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivation Enhanced BWL (Active Comparator): 12 week treatment program consisting of 2, 90-minute individual sessions with a focus on motivation, followed by weekly PDF modules via email, and reporting of key behaviors and feedback via email. Participants will pick from one of three dietary goals and one of three physical activity goals.
  Interventions: Behavioral: Motivation Enhanced BWL
- Brief Behavioral Weight Loss (BWL) (Active Comparator): 12 Week treatment program consisting of 2, 90-minute individual sessions, followed by weekly PDF modules via email, and reporting of key behaviors and feedback via email. Treatment consistent with behavioral weight loss, low calorie, low fat diet. Increased physical activity of up to 250 minutes/week.
  Interventions: Behavioral: Brief Behavioral Weight Loss (BWL)

INTERVENTIONS:
Behavioral: Brief Behavioral Weight Loss (BWL) — 12 Week treatment program consisting of 2, 90-minute individual sessions, followed by weekly PDF modules via email, and reporting of key behaviors and feedback via email. Treatment consistent with behavioral weight loss, low calorie, low fat diet. Increased physical activity of up to 250 minutes/week.
  Arms: Brief Behavioral Weight Loss (BWL)
Behavioral: Motivation Enhanced BWL — 12 week treatment program consisting of 2, 90-minute individual sessions with a focus on motivation, followed by weekly PDF modules via email, and reporting of key behaviors and feedback via email. Participants will pick from one of three dietary goals and one of three physical activity goals.
  Arms: Motivation Enhanced BWL

SUMMARY:
This study is a 2-arm randomized controlled trial to evaluate the feasibility, acceptability and preliminary efficacy of an MI-based program for weight loss in young adults.

DETAILED DESCRIPTION:
This study is a 2-arm randomized controlled trial to evaluate the feasibility, acceptability and preliminary efficacy of an MI-based program for weight loss in young adults. Participants will be assigned to either the MI Behavioral Weigh Loss or Behavioral Weight Loss arms - both arms will receive a 12-week Behavioral Weight Loss program, including 2 individual in-person sessions, followed by weekly Behavioral Weight Loss modules, reporting of key behaviors, and feedback on progress relative to goals, all via email. Session content will be quite distinct between the two arms, with an increased emphasis on personalized feedback relative to healthy norms, enhancing autonomous motivation, and choice surrounding diet and activity goals in the MIBWL arm. Assessments will take place at 0, and 3 months, followed by exit interviews to help refine the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-25 years of age.
* Body Mass Index (BMI) between 25 and 45 kg/m2.
* Men and women will be recruited.
* All race and ethnic groups will be recruited.

Exclusion Criteria:

1. Currently receiving treatment for Type 2 Diabetes, hypertension, hyperlipidemia, or report a history of cardiovascular disease.
2. Other health problems which may influence the ability to walk for physical activity or be associated with unintentional weight change, including cancer treatment within the past 5 years or tuberculosis.
3. Report a history of, or current diagnosed DSM-IV-TR eating disorder (i.e., anorexia nervosa or bulimia nervosa) or any current compensatory behaviors (e.g., vomiting, laxative use, excessive exercise).
4. Report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q). Individuals endorsing joint problems, prescription medication usage, or other medical conditions that could limit exercise will be required to obtain written physician consent to participate.
5. Report a history of any psychotic disorder, bipolar disorder, or organic brain syndromes; report hospitalization for any psychiatric disorder within the last 12 months.
6. Are currently participating in a weight loss program and/or taking weight loss medication.
7. Lost > 5% of body weight during the past 6 months or history of bariatric surgery.
8. Participation in any other research study that may interfere with this study.
9. Intend to move outside of the surrounding area within the time frame of the investigation or will be out of town / unavailable for three or more weeks during the initial intervention period.
10. Are pregnant, lactating, less than 6 months post-partum, or plan to become pregnant during the time frame of the investigation.
11. Failure to complete screening appointments. -

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Feasibility | 12 weeks
  Primary Aims Include:
  Primary Aim 1: To determine the feasibility of an MI-based approach to weight loss in young adults. Specifically, to demonstrate that we can: 1) recruit 18-25 year olds into the proposed program, 2) keep them engaged, as evidenced by achieving >80% attendance and >80% completion of tracking / reporting activities, and 3) retain them for assessments, as evidence by achieving >80% retention at 12 and 24 week visits.
Adherence | 12 weeks
  Primary Aim 2: To explore whether the MIBWL arm produces better adherence (see Aim 1, item 2), retention, autonomous motivation, and satisfaction, all of which may be related to better weight losses in the long-term.

SECONDARY OUTCOMES:
Weight Loss | 12 weeks
  To explore whether the MIBWL arm is a viable approach to weight loss in this age group. Specifically, within group, we will examine mean weight change and proportion of participants achieving a clinically significant weight loss (>5%). Although not powered to detect differences, we will also explore differences in mean weight change between the MIBWL and BBWL groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica G LaRose, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University School of Medicine, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No